CLINICAL TRIAL: NCT02941432
Title: Pilot Study of Effects and Tolerance of Black Tea Compress Treatment in Facial Eczema and Perioral Dermatitis
Brief Title: Black Tea Compresses for Facial Eczema and Perioral Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Iakov Shimanovich, MD, Attending Dermatologist, University of Luebeck
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Black Tea Trial
Record Dates: First submitted 2016-10-16; First posted 2016-10-21 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Eczema, Dermatitis
MeSH Terms: conditions — Eczema; Dermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Black tea (Other): Black tea compress treatment
  Interventions: Other: Black tea compress treatment

INTERVENTIONS:
Other: Black tea compress treatment — Wet compresses with black tea applied 4-5 times daily to the face for 6 days

SUMMARY:
Facial eczema and perioral dermatitis are clinical entities that develop exclusively in the face and present a special therapeutic challenge. Topical corticosteroids that are commonly applied to treat eczema/dermatitis at other body sites are best avoided in the face, as they may result in rapid atrophy of facial skin and in the long term rather aggravate facial dermatoses. Black tea compresses have been successfully used by German-speaking dermatologists to treat facial eczema/dermatitis for decades. The precise mechanism of action is unknown but is presumably based on astringent properties of tannins in the black tea and on the antiinflammatory action of a wet compress as such. This therapy is cheap, universally available and practically free of side-effects. Despite these perceived advantages the effects and tolerance of black tea compresses have not been formally studied to date. Therefore, the investigators plan to treat 25 patients with facial eczema/perioral dermatitis over a period of 6 days each within the current trial. The disease activity will be assessed before, during and after completion of treatment using several clinical scores. In addition, side-effects, if any, will be documented.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of facial eczema or perioral dermatitis
* minimum age of 18 years
* patient is capable of granting informed consent
* patient is expected to comply with the trial treatment protocol
* for outpatients: close place of residence

Exclusion Criteria:

* initiation or increase of systemic immunosuppressive or antibiotic treatment necessary
* psychiatric disease or other factors making poor patient compliance probable
* participation in another clinical trial within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-09-01; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Facial Eczema Activity and Severity Index (patients with facial eczema) | days 0, 3 and 6
Change in Perioral Dermatitis Severity Score (patients with perioral dermatitis) | days 0, 3 and 6
Change in Investigator´s Global Assessment Score (all patients) | days 0, 3 and 6
Change in Patient´s Self-Assessment Score (all patients) | days 0, 3 and 6
Change in Visual Analog Scale for pruritus in the face (patients with facial eczema) | days 0, 3 and 6
Change in Visual Analog Scale for tension feeling in the face (patients with perioral dermatitis) | days 0, 3 and 6

SECONDARY OUTCOMES:
Side-effects | days 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Iakov Shimanovich, MD, Principal Investigator — University of Lübeck
Locations (1):
- Department of Dermatology, University of Lübeck, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Yes
It is planned to publish the study results, including anonymized clinical patient data and photographs in a scientific journal.

REFERENCES:
- [Derived] Witte M, Krause L, Zillikens D, Shimanovich I. Black tea dressings - a rapidly effective treatment for facial dermatitis. J Dermatolog Treat. 2019 Dec;30(8):785-789. doi: 10.1080/09546634.2019.1573306. Epub 2019 Feb 3. PMID 30668184